CLINICAL TRIAL: NCT02874105
Title: Glenohumeral Re-centering During Closed Kinetic Chain for Shoulder Physiotherapy. A Prospective and Randomized Study.
Acronym: SCAPULEO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties for enrollment
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PO16022*
Record Dates: First submitted 2016-08-11; First posted 2016-08-22 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Subacromial Impingement of the Shoulder
Keywords: Medical treatment; physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- experimental group (Experimental): Dynamic Humeral Centering
  Interventions: Other: Group S: physiotherapy protocol with Dynamic Humeral Centering.
- control group (Active Comparator): Conventional physiotherapy
  Interventions: Other: Group C: physiotherapy protocol with Conventional physiotherapy.

INTERVENTIONS:
Other: Group C: physiotherapy protocol with Conventional physiotherapy.
  Arms: control group
Other: Group S: physiotherapy protocol with Dynamic Humeral Centering.
  Arms: experimental group

SUMMARY:
The rotator cuff tendinopathy is very common and associated with degenerative or traumatic changes of the rotator cuff and/or the sub-acromial bursa or the long head of the biceps. Lesions go of the simple tendinopathy without tear to the full-thickness tear of the cuff which means a loss of mobility or strength. The origin of this pathology remains controversial and many causes have been evoked (subacromial mechanical impingement, degenerative changes, muscle imbalance…). The clinical impairment is not always the same and varies from a painful shoulder with correct range of motion to a pseudoparalysis shoulder. The first treatment of the rotator cuff pathology is always non surgical and consists in relative resting, painkillers and/or non-steroidal anti-inflammatory drugs (NSAD) and physiotherapy. The aim of this management is to relieve pain and to restore the mobility and a good function of the shoulder.

There is no consensus about the physiotherapy protocol for the treatment of the rotator cuff tendinopathy. In France, the most used physiotherapy protocol uses the strengthening of the muscles which stabilize the scapula (rhomboide muscles, trapezius and serratus anterior) and which lower the humerus (pectoralis major, latissimus dorsi and teres major). The aim of this approach is to augment the subacromial space in order to decrease the inflammation of the rotator cuff tendons and the associated pain. A technique of Dynamic Humeral Centering (DHC) uses a new method of glenohumeral centering in closed kinetic chain has been described ("3C Concept" for Centering in a Closed Chain). Dynamic humeral centring (DHC) is a modality of physiotherapy that aims to prevent subacromial impingement of rotator cuff tendons. In order to simplify and to improve its reliability, a special device called Scapuleo® has been developed. The aim of this device is to help the physiotherapist to realize simultaneously a subacromial decompression, a specific strengthening of the rotator cuff muscles and an optimal activation of the lower trapezius and the anterior serratus.

Our hypothesis was that the DHC was not inferior to the conventional physiotherapy protocol for the medical treatment of the rotator cuff tendinopathy without full-thickness tear.

We proposed a prospective and randomized study. All the patients treated in our department for simple tendinopathy of the rotator cuff or partial thickness tear were included in this study after signed consent. The physiotherapy protocol consists in 20 sessions of either "Conventional program" (Control group) or "Dynamic Humeral Centering" (Study group). The clinical evaluation included the range of motion measurement, Constant Score, Quick-DASH and Oxford Shoulder Score at 3 months and 6 months. Patients were blinded to the study hypothesis. The assessor of all outcomes was blinded to the interventions.

DETAILED DESCRIPTION:
Shoulder impingement accounts for 44 to 65% of shoulder complaints during physician visits. Shoulder impingement has been classified into two main categories: structural and functional. The structural impingement can be caused by narrowing of the subacromial space resulting from a reduction in the space due to bony growth or soft-tissue inflammation. The functional impingement or superior migration of the humeral head can be caused by weakness and/or muscle imbalance. It is possible that some subacromial impingement results from a combination of both structural and functional factors. Subacromial impingement occurs when the structures in the SAS (rotator cuff, biceps tendon long head, and subacromial bursa) become compressed and inflamed under the coracoacromial ligament. The suprasinatus tendon in particular is at highest risk for irritation and subsequent injury because it is the most likely to contact the acromion when the humerus is abducted to 90° and internally rotated 45°.

The clinical impairment is not always the same and varies from a painful shoulder with correct range of motion to a pseudoparalysis shoulder. The first treatment of this subacromial impingement is always non surgical and consists in relative resting, painkillers and/or non-steroidal anti-inflammatory drugs (NSAD) and physiotherapy. The aim of this treatment is to relieve pain and to restore the mobility and a good function of the shoulder.

There is no consensus about the physiotherapy protocol for the treatment of the shoulder impingement. In France, the most used physiotherapy protocol uses the strengthening of the muscles which stabilize the scapula (rhomboide muscles, trapezius and serratus anterior) and which lower the humerus (pectoralis major, latissimus dorsi and teres major). The aim of this approach is to augment the subacromial space in order to decrease the inflammation of the rotator cuff tendons and the associated pain. A technique of Dynamic Humeral Centering (DHC) uses a new method of glenohumeral centering in closed kinetic chain has been described ("3C Concept" for Centering in a Closed Chain). Dynamic humeral centring (DHC) is a modality of physiotherapy that aims to prevent subacromial impingement of rotator cuff tendons. In order to simplify and to improve its reliability, a special device called Scapuleo® has been developed. The aim of this device is to help the physiotherapist to realize simultaneously a subacromial decompression, a specific strengthening of the rotator cuff muscles and an optimal activation of the lower trapezius and the anterior serratus.

Our hypothesis was that the DHC was not inferior to the conventional physiotherapy protocol for the medical treatment of the subacromial impingement.

We proposed a prospective and randomized study. All the patients treated in our department for simple tendinopathy of the rotator cuff or partial thickness tear were included in this study after signed consent. The physiotherapy protocol consisted in 20 sessions of either "Conventional program" (Control group) or "Dynamic Humeral Centering" (Study group). The clinical evaluation included the range of motion measurement, Constant Score, Quick-DASH and Oxford Shoulder Score at 3 months and 6 months. Patients were blinded to the study hypothesis. The assessor of all outcomes was blinded to the interventions.

The rhythm of the physiotherapy sessions was the same in both groups (3 sessions per week for 3 weeks, 2 sessions per week for 3 weeks and 1 session per week for 5 weeks). All patients received passive mobilization of the shoulder without pain and muscle stretching. Each physiotherapy session lasted 30 minutes and included massage or hot physiotherapy in case of VAS (visual analogic scale) of pain superior to 6/10.

ELIGIBILITY:
Inclusion Criteria:

* Painful shoulder causes by tendinopathy of the rotator cuff (without full-thickness tear)
* Diagnosis based on a MRI (dating less than 6 months)

Exclusion Criteria:

* Tendinopathy of the rotator cuff with full-thickness tear
* Stiffness of the shoulder (loss of more than 20° in passive external rotation or passive forward elevation)
* Previous shoulder surgery (less than 12 months)
* Previous subacromial injection (less than 6 months)
* Context of worker's compensation claims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Functional status of the shoulder | 6 months
  Functional status of the shoulder evaluated using the Constant & Murley Score

SECONDARY OUTCOMES:
Functional status of the shoulder | 3 months
  Functional status of the shoulder evaluated using the Constant & Murley Score
Disabilities of the Arm, Shoulder and Hand score | 3 months
  Disabilities of the Arm, Shoulder and Hand score evaluated using the Quick-DASH (short form), self reported questionnaire (12 questions)
Disabilities of the Arm, Shoulder and Hand score | 6 months
  Disabilities of the Arm, Shoulder and Hand score evaluated using the Quick-DASH (short form), self reported questionnaire (12 questions)
Functional status of the shoulder | 3 months
  Functional status of the shoulder evaluated using Oxford Shoulder Score, self reported questionnaire (12 questions)
Functional status of the shoulder | 6 months
  Functional status of the shoulder evaluated using Oxford Shoulder Score, self reported questionnaire (12 questions)
pain | 3 months
  Shoulder pain evaluated using a visual analogic pain scale
pain | 6 months
  Shoulder pain evaluated using a visual analogic pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France